CLINICAL TRIAL: NCT02488629
Title: An Open-Label, Phase II Study to Evaluate SCB01A in Patients With Recurrent or Metastatic Squamous Cell Head and Neck Cancer Who Have Received Platinum-Based Treatment
Brief Title: Study of SCB01A in Patient With Head and Neck Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SynCore Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCB01A-21
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Results first posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Head and Neck Squamous Cell Carcinoma
Keywords: Head and neck squamous cell carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SCB01A (Experimental): This study is a single arm, open-label, Phase II trial
  Interventions: Drug: SCB01A

INTERVENTIONS:
Drug: SCB01A — This study is a single arm, open-label, Phase II trial

SUMMARY:
To evaluate the safety and efficacy of SCB01A in head and neck cancer.

DETAILED DESCRIPTION:
The study is designed to evaluate the safety and efficacy of SCB01A in patients with recurrent or metastatic squamous cell carcinoma in head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed squamous cell carcinoma of head and neck
2. Patients with nonresectable, unfeasible radiotherapy, recurrent or metastatic carcinoma, after previous treatment with platinum agent.
3. At least one measurable tumor lesion according to RECIST
4. Suitable Eastern Cooperative Oncology Group (ECOG) performance status
5. All eligible patients of childbearing potential have to use effective contraception
6. Signed informed consent before enrolment

Exclusion Criteria:

1. Receiving Chemotherapy, radiation therapy, major surgery or investigational agents
2. Severe pulmonary obstructive or restrictive disease
3. Uncontrolled inflammatory disease
4. Clinically significant cardiac disease
5. Results of laboratory tests
6. Pregnancy or nursing status
7. Known hypersensitivity to any component of SCB01A
8. History of exposure to SCB01A or its analogues
9. History of malignancy other than head and neck cancer
10. History of active or significant neurological disorder or psychiatric disorder
11. Any other reason the investigator deems the patient to be unsuitable for the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hung Wang, MSc, Study Director — SynCore Biotechnology Co., Ltd.
Locations (5):
- Taiwan (5):
  - Keelung Chang Gung Memorial Hospital & lovers lake branch, Keelung
  - National Cheng Kung University Hospital, Tainan
  - MacKay Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: No subjects were enrolled in Run-in Phase I: Dose 3 (18 mg/m²), Dose 4 (24 mg/m²), and Phase II.
Groups:
- SCB01A 3.25 mg/m²: Three subjects (expanded to six subjects in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 3.25 mg/m² (Dose 1) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 1).
- SCB01A 12 mg/m²: Three subjects (expanded to six subjects in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 12 mg/m² (Dose 2) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 2).
- SCB01A 18 mg/m²: Three subjects (expanded to six subjects in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 18 mg/m² (Dose 3) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 3).
- SCB01A 24 mg/m²: Three subjects (expanded to six subjects in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 24 mg/m² (Dose 4) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 4).
Period: Overall Study
Arm/Group | SCB01A 3.25 mg/m² | SCB01A 12 mg/m² | SCB01A 18 mg/m² | SCB01A 24 mg/m²
Started | 3 | 2 | 0 | 0
Completed | 0 (All 5 patients withdrew from the study. The reasons for premature study discontinuation were RECIST disease progression (4 patients [80%]) and voluntary discontinuation (1 [20%]). All 5 patients were enrolled in the Run-in Phase I and no patients were enrolled in Phase II.) | 0 | 0 | 0
Not Completed | 3 | 2 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1); Run-in Phase I (Dose Escalation Phase): 12 mg/m² (Dose 2): Run-in Phase I (Dose Escalation Phase):
  The first part of the study involved dose-escalation, in which successive cohorts of 3 patients (expanded to 6 patients in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 3.25 mg/m² (Dose 1) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 1) until 24 mg/m² (3.25→12→18→24). Dose escalation assessment was based on tolerability observed during 3 cycles of treatment.
- Total: Total of all reporting groups
Arm/Group | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1) | Run-in Phase I (Dose Escalation Phase): 12 mg/m² (Dose 2) | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 56.3 [56 to 57] | 53.5 [52 to 55] | 55.2 [52 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 3 | 2 | 5
ECOG at Screening visit [Count of Participants; unit: Participants] — Measure Description:
  ECOG 0: Fully active, able to carry on all pre-disease performance without restriction.
  ECOG 1: Restricted in physically strenous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  ECOG 2: Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours. Population: Data not collected for 12 mg/m² (Dose 2) cohort as the 2 subjects from the Dose 2 did not complete 3 treatment cycles.
  Participants
    number analyzed (Participants) | 3 | 0 | 3
    0 | 0 |  | 0
    1 | 2 |  | 2
    2 | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Disease Control Rate (DCR)
Description: To assess the DCR (=complete response (CR) + partial response (PR) + stable disease (SD)) at the end of the 9th week (3 cycles, each cycle consisted of 21 days) after treatment with SCB01A, according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sumdiameterswhile on study.
Time Frame: 9 weeks from 1st administrationm drug
Population: Data not collected for 12 mg/m² (Dose 2) cohort as the 2 subjects from the Dose 2 did not complete 3 treatment cycles.
Measure: Count of Participants; unit: Participants
Groups:
- Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1): The first part of the study involved dose-escalation, in which successive cohorts of 3 patients (expanded to 6 patients in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 3.25 mg/m² (Dose 1) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 1) until 24 mg/m² (3.25→12→18→24).
Arm/Group | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1)
Number analyzed (Participants) | 3
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 0
  Stable Disease (SD) | 1
  Progressive Disease (PD) | 2

2. Secondary Outcome: To Assess the Overall Survival Rate
Description: To assess the overall survival (OS) rate at 36 weeks after first treatment with SCB01A in patients with recurrent or metastatic squamous cell head and neck cancer who have previously been treated with platinum therapy.
Time Frame: an expected average of 36 weeks
Population: Data not collected for 12 mg/m² (Dose 2) cohort as the 2 subjects from the Dose 2 did not complete 3 treatment cycles.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1)
Number analyzed (Participants) | 3
weeks | 25.57 [10.14 to 32.14]

3. Secondary Outcome: To Assess the Progression-free Survival According to RECIST v.1.1
Description: RECIST v.1.1: Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: an expected average of 12 weeks
Population: Data not collected for 12 mg/m² (Dose 2) cohort as the 2 subjects from the Dose 2 did not complete 3 treatment cycles.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1)
Number analyzed (Participants) | 3
weeks | 8.71 [8.43 to 12.14]

ADVERSE EVENTS:
Time Frame: From the time of informed consent obtained until 28 days after the last dose of study treatment
Groups:
- Run-in Phase I (Dose Escalation Phase): 12 mg/m² (Dose 2): The first part of the study involved dose-escalation, in which successive cohorts of 3 patients (expanded to 6 patients in the event of a dose-limiting toxicity) were enrolled and administered 3 cycles of i.v. SCB01A at a dose of 3.25 mg/m² (Dose 1) on Days 1 and 8 of each cycle in a 3-week cycle (Dose 1) until 24 mg/m² (3.25→12→18→24).
Arm/Group | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1) | Run-in Phase I (Dose Escalation Phase): 12 mg/m² (Dose 2)
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1) (N=3) | Run-in Phase I (Dose Escalation Phase): 12 mg/m² (Dose 2) (N=2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Phase I (Dose Escalation Phase): 3.25 mg/m² (Dose 1) (N=3) | Run-in Phase I (Dose Escalation Phase): 12 mg/m² (Dose 2) (N=2)
Facial pain (General disorders) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (2) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (3) | 0 (0)
Feeling cold (General disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Tinea manuum (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Salivary gland pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 0 (0) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2016-07-25): https://cdn.clinicaltrials.gov/large-docs/29/NCT02488629/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT02488629/SAP_001.pdf